CLINICAL TRIAL: NCT03538080
Title: Evaluation du pré-marquage Par AccuVein® au Cours Des échographies Doppler de repérage saphène.
Brief Title: ACCUvein Measure Before ULtrasound as A facilitataTION Tool for Venous Marking
Acronym: ACCUMULATION
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2018-A01101-54
Record Dates: First submitted 2018-01-18; First posted 2018-05-25 (Actual); Last update posted 2020-08-14 (Actual); Status verified 2020-08

CONDITIONS: Other Diseases of Veins and Lymphatics
Keywords: venous disease; peripheral vascular disease; vascular surgery; ultrasound imaging
MeSH Terms: conditions — Peripheral Vascular Diseases | interventions — Ultrasonography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ACCUVEIN plus ultrasound (Experimental): Patients referred for marking of saphenous veins before varicose vein surgery or for saphenectomy for vascular or coronary artery bypass grafting will have marking with Accuvein and ultrasound
  Interventions: Device: ACCUVEIN plus ultrasound
- Ultrasound only (Sham Comparator): Patients referred for marking of saphenous veins before varicose vein surgery or for saphenectomy for vascular or coronary artery bypass grafting will have marking with ultrasound only.
  Interventions: Device: Ultrasound only

INTERVENTIONS:
Device: ACCUVEIN plus ultrasound — Intervention is marking of the saphenous veins with ACCUVEIN system. The AccuVein® AV400 vein illumination system is a laser imaging system that detects superficial veins up to 10 mm deep and digitally displays, through a projected red light, a map of the vascularization on the surface of the skin. in real time, allowing clinicians to check vein permeability and position.
  This system is portable and lightweight. It can be easily cleaned, and requires no calibration or adjustment. It does not require any contact with the patient. Second time is completion of marking by ultrasound if necessary
  Arms: ACCUVEIN plus ultrasound
Device: Ultrasound only — Intervention is marking with ultrasound imaging as in usual practice.
  Arms: Ultrasound only

SUMMARY:
Ultrasound marking of saphenous veins before varicose vein surgery or for saphenectomy for vascular or coronary artery bypass grafting is a long, tedious, low-grading examination, generating overconsumption of many consumables including marking markers that may damage the probes, of the modern and expensive ultrasound doppler. Augmented reality devices can visualize the superficial veins and hope to simplify the investigation, improve the comfort of the patient during the examination by significantly reducing the time of the examination. There is few data in the literature on the value of using augmented reality devices of this type. The AccuVein® system is a patient-friendly, non-contact, non-invasive technique that minimizes discomfort due to standing time and thus improves patient comfort.

DETAILED DESCRIPTION:
At admission eligible patients are proposed to participate. Written consent is signed after complete oral and written explanation of the protocol is signed. No register of non-included patients will be kept. In included patients, in parallel to the standard ultrasound investigation for marking of saphenous veins for which the patient is referred, AccuVein® system will be performed as explained later in arm description.

Usual ongoing treatments are obtained by history and recorded. The end of the visit is the end of the participation of the subjects.

ELIGIBILITY:
Inclusion Criteria:

* Patients referred for venous marking
* Affiliation to the French National healthcare system
* French speaking patients

Exclusion Criteria:

* pregnancy
* inability to understand the study goal
* patients protected by decision of law

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2018-09-03 (Actual); Primary Completion 2019-06-20 (Actual); Study Completion 2019-06-20 (Actual)

PRIMARY OUTCOMES:
Time to perform the saphenous vein marking with AccuVein® system | inclusion
  Time to perform the marking of the leg (from the beginning of marking until the end of marking of the leg concerned), using the AccuVein® system supplemented by a ultrasound doppler , compared to the ultrasound doppler reference technique.

SECONDARY OUTCOMES:
Degree of satisfaction of the vascular physician and the surgeon | inclusion
  Likert scale of satisfaction of the surgeon and the vascular physician, according to the use of AccuVein® or the ultrasound doppler reference technique for the identification of saphenous veins
Rate of consumables | inclusion
  Number of marker pens needed during marking, according to the use of AccuVein® or the ultrasound doppler reference technique for the detection of saphenous veins

CONTACTS AND LOCATIONS:
Overall Officials: HENNI MD SAMIR, PhD, Principal Investigator — UH Angers
Locations (1):
- UH Angers, Angers, France